CLINICAL TRIAL: NCT02944461
Title: Efficacy and Safety of Aczone 7.5% Gel in the Treatment of Truncal Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACZ1601
Record Dates: First submitted 2016-10-04; First posted 2016-10-25 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapsone gel 7.5% (Experimental): Dapsone gel 7.5% to be applied to truncal acne once daily for 16 weeks.
  Interventions: Drug: Dapsone 7.5 % gel

INTERVENTIONS:
Drug: Dapsone 7.5 % gel — Dapsone gel 7.5% applied once daily to truncal acne
  Other Names: Aczone

SUMMARY:
To determine if Dapsone (Aczone) 7.5% gel is a safe and effective treatment for acne on the trunk

DETAILED DESCRIPTION:
This is an open label pilot study to determine the safety and efficacy of Dapsone (Aczone) 7.5% gel applied daily to the trunk for acne. Subjects will apply Dapsone for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any race and at least 12 years of age.
* Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline and practice a reliable method of contraception throughout the study.
* Truncal acne IGA score of 3.
* Able to understand the requirements of study and sign Informed Consent/HIPAA forms.

Exclusion Criteria:

* Female subjects who are pregnant , breast feeding or are of childbearing potential who are not willing to use a reliable method birth control.
* Subjects who have an allergy or sensitivity to any component of the test medication.
* Subjects who have not complied with the proper wash out periods for prohibited medications.
* Evidence of recent drug or alcohol abuse.
* Skin disease /disorder that might interfere with the diagnosis or evaluation of truncal acne.
* Exposure to an investigational drug within 30 days of the Baseline visit.
* Medical condition that contraindicates the subject's participation in the study.
* History of poor cooperation, non-compliance with medical treatment or unreliability.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Study Director — DermResearch PLLC
Locations (3):
- United States (3):
  - Dermatology and Laser Surgery, Sacramento, California
  - DermResearch, PLLC, Louisville, Kentucky
  - James Q. DelRosso DO, LLC, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapsone Gel 7.5%
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dapsone Gel 7.5%
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Achieve at Least a Two Grade Improvement and a Rating of Clear or Almost Clear on the Investigator Global Assessment (IGA) Scale
Description: Investigator will evaluate global acne severity using the IGA scale as follows: 1= Clear Skin, 2 = Almost Clear, 3 = Mild Severity, 4 = Severe, 5 = Very Severe
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapsone Gel 7.5%
Number analyzed (Participants) | 15
Participants
  week 4 | 0
  week 10 | 3
  week 16 | 7

2. Secondary Outcome: The Percent Change in Inflammatory Lesion Count at Week 16 Compared to Baseline
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Arm/Group | Dapsone Gel 7.5%
Number analyzed (Participants) | 15
percent change in lesion count | -74 (21)

3. Secondary Outcome: The Percent Change in Non-inflammatory Lesion Count at Week 16 Compared to Baseline
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Arm/Group | Dapsone Gel 7.5%
Number analyzed (Participants) | 15
percent change in lesion count | -72 (28)

4. Secondary Outcome: The Percent Change in Total Lesion Count at Week 16 Compared to Baseline
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Arm/Group | Dapsone Gel 7.5%
Number analyzed (Participants) | 15
percent change in lesion count | -73 (23)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Dapsone Gel 7.5%
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapsone Gel 7.5% (N=20)
infected abrasions of legs (Skin and subcutaneous tissue disorders) | 1 (1)
gum graft surgery (Surgical and medical procedures) | 1 (1)
stye, right eye (Eye disorders) | 1 (1)
sunburn arms/chest/back (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02944461/Prot_SAP_000.pdf